CLINICAL TRIAL: NCT02618135
Title: Effectiveness of a Brain-Computer Interface-based Programme for the Treatment of Autism Spectrum Disorder and Attention Deficit Hyperactivity Disorder in Children: A Pilot Study
Brief Title: Brain-Computer Interface-based Programme for the Treatment of ASD/ADHD
Acronym: ASDBCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Institute of Mental Health, Singapore (Other); Agency for Science, Technology and Research (Other)
Responsible Party: Principal Investigator, Lee Tih Shih, Associate Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/00841
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): 10 child participants in the intervention group will take part in a total of 24 sessions spread over an 8-week period, and a final follow-up review 1 month after the completion of the training session. If sessions are missed during the 8-weeks period due to unforeseen circumstances (e.g. sickness, travel plans), arrangements will be made for participants to attend up to 5 BCI-based therapy sessions per week. All participants will have to complete a minimum of 20 sessions within the 8-weeks period for treatment efficacy.
  Interventions: Other: Intervention Group
- Control Group (Other): 10 child participants in the control group will not receive BCI training during the first 8 weeks of their study participation; they will act as controls. At week 9, subjects in this group will go through the BCI training similar to the intervention group. If sessions are missed during the 8-weeks period due to unforeseen circumstances (e.g. sickness, travel plans), arrangements will be made for participants to attend up to 5 BCI-based therapy sessions per week. All participants will have to complete a minimum of 20 sessions within the 8-weeks period for treatment efficacy. They will take part in a total of 24 sessions spread over an 8-week period, followed by a final follow-up review 1 month after the completion of the training sessions.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Intervention Group — Each participant will first need to master a simple concentration task before moving on to play a series of training tasks. An eye gaze tracker connected to the computer will detect the location of eye gaze on the computer screen. The game progresses according to how well the participant can focus their eye gaze on correct objects and sustain their attention. Each task employs the BCI system, and is controlled by the child's concentration. As the child attends to activities on a computer screen, their EEG waves will be recorded simultaneously via the EEG sensors through Bluetooth technology.
  Other Names: BCI Training
  Arms: Intervention Group
Other: Control Group — Participants will wait for 8 weeks before training intervention begins.
  Each participant will first need to master a simple concentration task before moving on to play a series of training tasks. An eye gaze tracker connected to the computer will detect the location of eye gaze on the computer screen. The game progresses according to how well the participant can focus their eye gaze on correct objects and sustain their attention. Each task employs the BCI system, and is controlled by the child's concentration. As the child attends to activities on a computer screen, their EEG waves will be recorded simultaneously via the EEG sensors through Bluetooth technology.
  Other Names: Waitlist BCI Training
  Arms: Control Group

SUMMARY:
This project involves creating a novel and personalised BCI training system that targets social and communication difficulties, and inattentive symptoms problems often found in ASD/ADHD children. 20 participants between the age of 8 and 12 will be recruited and they will undergo 24 training sessions over an 8-week period. During these sessions, the children will play a computer game interface specifically designed to train attention and facial and emotional recognition, while using our BCI device. To further reinforce the treatment, the training system has been enhanced with the inclusion of an eye-tracker to target the lack of preferential eye contact that children with ASD exhibit. The investigators hypothesize that participants will show improvements in social skills and attention post treatment.

DETAILED DESCRIPTION:
This pilot trial aims to improve attention levels in children with comorbid ASD/ADHD. Twenty participants aged 8 to 12 years with comorbid ASD/ADHD will be recruited. Most therapy involves at least a total of 20 sessions (4); as such, the intervention protocol includes 24 sessions followed by a follow up one month after completion. The participants will attend 24 brain training sessions over an 8-week period, playing computer games designed for improving attention, facial recognition, and emotion recognition.

Participants will be randomized to either the Intervention or Waitlist-Control study arm group, where the latter proceeds with training only after a wait-time of 8 weeks. The investigators hypothesize that participants in the Intervention group will show improved symptoms compared to the Waitlist-Control group at week 8. This pilot study will provide preliminary data to support the efficacy of the investigators new BCI-based training programme and potentially pave the way for a larger randomized controlled trial.

Children with comorbid ASD/ADHD have greater impairments in attention, social skills and eye gaze. The investigators believe that focusing on these symptoms might lead to potentially better treatment outcomes. Also, current treatments for ASD/ADHD are limited in that they are taxing, time-consuming, and incur side effects. If the BCI-based training programme has a positive impact on children diagnosed with ASD and ADHD, it can potentially be an alternative long-term treatment. Unlike medications and behavioural interventions, neurofeedback therapy has no side effects and may be more engaging for children. It has the potential to be made available eventually for use at the patient's own home and can therefore be administered at one's own time and convenience.

In 2010, the PI and his team conducted a pilot study to investigate a novel intervention for treatment of ADHD. The study involved subjects 7 to 12 years of age diagnosed with either combined or inattentive ADHD subtypes. The subjects received 20 sessions of BCI training over a 10-week period. The BCI training is an innovative design integrating neurofeedback system using an algorithm to analyze EEG brain waves, using it to drive a computer interface by sustaining a certain threshold of attention. Teachers of children in the intervention group reported larger improvements in the ADHD inattentive score although this was not statistically significant. Parents also fed back that the intervention was relatively safe to use and free of adverse effects.

In 2012, the team completed another study that improved upon the technology and investigated the feasibility of the new training programme (with a simpler headset using two dry lead sensors instead of an EEG cap) on 20 unmedicated ADHD children participants. The treatment intervention was intensified to 24 sessions over 8 weeks followed by 3 monthly booster training sessions. An additional component was added to the training module where participants were required to complete a stroop task calibration process before the training. This is to personalise the intervention and improve accuracy of the EEG parameters. In this open-label trial, parents reported statistically significant improvements in both inattentive and hyperactive-impulsive symptoms on the ADHD Rating Scale at 8 weeks, which further suggests the potential efficaciousness of the novel BCI-based training programme as a potentially efficacious treatment for ADHD.

In 2013, a larger-scale randomised controlled trial began to further investigate the efficacy of the BCI training on treating inattentive symptoms of ADHD. The randomized study aims to enroll 160 children between the age of 6 to 12 who will undergo 24 sessions of BCI training sessions over 8 weeks followed by 3 booster sessions. ADHD symptoms will be assessed primarily by blinded clinicians and parents as well as based on feedback obtained from respective school teachers. The study is currently ongoing and is estimated to complete by July 2016. Therapy using non-invasive BCI system-based games may represent an alternative treatment for children with ADHD and ASD. If demonstrated to be efficacious, parents are likely to prefer this as compared to current treatment modalities of medications (with potentially serious side effects) and behavior management (parents generally find this difficult and challenging). Children themselves are also more likely to enjoy the treatment and hence, comply better.

In the longer term, this approach and system may have potential for attention and cognitive enhancement for patients with cognitive impairment or early dementia.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for ASD, based on Autism Diagnostic Observation Scale (ADOS) and/or Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM IV-TR) / 5th edition (DSM 5);
* Meets diagnostic criteria for ADHD inattentive or combined subtype, based on the Computerised Diagnostic Interview for Children (C-DISC);
* Score 12 and above on the ADHD Rating Scale (ADHD-RS);
* IQ above 70;
* If on medication, dose has been stable or unchanged for at least preceding 3 months
* Parents and teachers are English-speaking

Exclusion Criteria:

1. Co-morbid severe psychiatric condition or known sensory-neural deficit e.g. complete blindness or deafness.
2. Color blindness
3. History of epileptic seizures.
4. Known to have developmental delay (i.e. IQ 70 and below).
5. Predominantly hyperactive/impulsive subtype of ADHD.
6. Change in dosage of medication (if on medication)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
ADHD Rating Scale (clinicians) | Week 1 to Week 8
  The primary outcome of this study will be the change in the inattentive score on the ADHD Rating Scale as rated by the clinicians from week 1 to week 8.

SECONDARY OUTCOMES:
ADHD Rating Scale (parent) | Week 1 to Week 8
  The change in the inattentive score of the ADHD RS rated by parent from week 1 to week 8.
ADHD Rating Scale (clinician and parent) | Week 1 to Week 8
  The change in the inattentive score of the ADHD RS rated by clinician and parent from week 1 to week 8.
ADHD Rating Scale | Week 1 to Week 8
  The change in parent rated ADHD-RS from week 1 to week 8.
Social Responsiveness Scale | Week 1 to Week 8
  The change in parent rated SRS from week 1 to week 8.
Clinical Global Assessment Scale (C-GAS) | Week 1 to Week 8
  The change in clinician rated CGAS and CGI scores from week 1 to week 8.
Clinical Global Impression Severity Scale (CGI-S) | Week 1 to Week 8
  The change in clinician rated CGAS and CGI scores from week 1 to week 8.
Clinical Global Impression Improvement Scale (CGI-I) | Week 1 to Week 8
  The change in clinician rated CGAS and CGI scores from week 1 to week 8.
Conners' Continuous Performance Test (CPT-II) | Week 1 to Week 8

OTHER OUTCOMES:
Pediatric Adverse Event Rating Scale (PAERS) | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Choon Guan Lim, Principal Investigator — Institute of Mental Health, Singapore
Locations (1):
- Institute of Mental Health, Singapore, Singapore

REFERENCES:
- [Background] Jang J, Matson JL, Williams LW, Tureck K, Goldin RL, Cervantes PE. RETRACTED: Rates of comorbid symptoms in children with ASD, ADHD, and comorbid ASD and ADHD. Res Dev Disabil. 2013 Aug;34(8):2369-78. doi: 10.1016/j.ridd.2013.04.021. Epub 2013 May 22. PMID 23708709
- [Background] Rommelse NN, Franke B, Geurts HM, Hartman CA, Buitelaar JK. Shared heritability of attention-deficit/hyperactivity disorder and autism spectrum disorder. Eur Child Adolesc Psychiatry. 2010 Mar;19(3):281-95. doi: 10.1007/s00787-010-0092-x. Epub 2010 Feb 11. PMID 20148275
- [Background] Coben R, Linden M, Myers TE. Neurofeedback for autistic spectrum disorder: a review of the literature. Appl Psychophysiol Biofeedback. 2010 Mar;35(1):83-105. doi: 10.1007/s10484-009-9117-y. PMID 19856096
- [Background] Linden M, Habib T, Radojevic V. A controlled study of the effects of EEG biofeedback on cognition and behavior of children with attention deficit disorder and learning disabilities. Biofeedback Self Regul. 1996 Mar;21(1):35-49. doi: 10.1007/BF02214148. PMID 8833315
- [Background] Gevensleben H, Holl B, Albrecht B, Vogel C, Schlamp D, Kratz O, Studer P, Rothenberger A, Moll GH, Heinrich H. Is neurofeedback an efficacious treatment for ADHD? A randomised controlled clinical trial. J Child Psychol Psychiatry. 2009 Jul;50(7):780-9. doi: 10.1111/j.1469-7610.2008.02033.x. Epub 2009 Jan 12. PMID 19207632
- [Background] Lim CG, Lee TS, Guan C, Sheng Fung DS, Cheung YB, Teng SS, Zhang H, Krishnan KR. Effectiveness of a brain-computer interface based programme for the treatment of ADHD: a pilot study. Psychopharmacol Bull. 2010;43(1):73-82. PMID 20581801
- [Background] Lee TS, Goh SJ, Quek SY, Phillips R, Guan C, Cheung YB, Feng L, Teng SS, Wang CC, Chin ZY, Zhang H, Ng TP, Lee J, Keefe R, Krishnan KR. A brain-computer interface based cognitive training system for healthy elderly: a randomized control pilot study for usability and preliminary efficacy. PLoS One. 2013 Nov 18;8(11):e79419. doi: 10.1371/journal.pone.0079419. eCollection 2013. PMID 24260218
- [Background] Jones W, Carr K, Klin A. Absence of preferential looking to the eyes of approaching adults predicts level of social disability in 2-year-old toddlers with autism spectrum disorder. Arch Gen Psychiatry. 2008 Aug;65(8):946-54. doi: 10.1001/archpsyc.65.8.946. PMID 18678799